CLINICAL TRIAL: NCT04321850
Title: Impact of the Use of Zinc in the Prevention of Oral Mucositis in Pediatric Patients With Lymphoblastic Acute Leukemia.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Health restrictions due to the COVID-19 pandemic
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Marta Zapata Tarrés, Pediatrician oncologist, National Institute of Pediatrics, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 036/2019
Record Dates: First submitted 2020-03-07; First posted 2020-03-25 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Oral Mucositis
Keywords: Zinc; Leukemia, Acute Lymphoblastic
MeSH Terms: conditions — Stomatitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Zinc Sulfate; Zinc; Mannitol

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized to designate them in the control group (Group1 placebo) or intervention group (Group 2 zinc). The zinc / placebo intervention will be administered orally in tablets of 50-100 mg / day, from day 1 of chemotherapy until the end of the consolidation phase (2 to 2.5 months).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient and the investigator will be blinded; for this, the 50 mg zinc and placebo tablets will be similar in size, color, shape, weight and taste; the bottles will be classified into codes A and B, which in turn will have the same shape, size and color. All of the above will be done through the Pharmaceuticals GREMAR S.A. de C.V., which is a Mexican company that has a line of food supplements located in Mexico City.
  An independent investigator (who will be blinded for the purpose of the study) will be requested to receive the medications (zinc / placebo) prepared by the Pharmaceuticals GREMAR S.A. of C.V., so that it provides to the principal investigator only the bottles coded as "A" and "B". At the end of the intervention, the independent investigator will be asked to reveal the coding of the medications to determine which group (Group 1 placebo or Group 2 zinc) corresponds to treatment A and B respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Placebo Comparator): Control
  Interventions: Drug: Placebo oral tablet
- Group 2 (Experimental): Intervention (Zinc)
  Interventions: Drug: Zinc Sulfate 50 Mg Tab

INTERVENTIONS:
Drug: Zinc Sulfate 50 Mg Tab — The tablets were manufactured specifically for this study.
  Other Names: Zinc
  Arms: Group 2
Drug: Placebo oral tablet — The tablets were manufactured specifically for this study.
  Other Names: Manitol
  Arms: Group1

SUMMARY:
Oral mucositis (OM) is a secondary complication of chemo/radiotherapy, which causes pain, dysphagia and predisposition to infections, being a frequent reason for hospitalization that may have an impact on the prognosis of cancer patients. Various interventions for the prevention of OM have been studied, including the use of zinc, which is a micronutrient that participates in various cellular functions and in wound repair, while showing a reduction in the incidence and severity of MO, so the purpose of the present study is to evaluate the impact of the use of zinc in the prevention of oropharyngeal mucositis in pediatric patients with acute lymphoblastic leukemia in chemotherapy, comparing it with the use of placebo.

Hypothesis: The use of zinc reduces the incidence and severity of OM in pediatric patients with ALL in chemotherapy compared to the control group.

DETAILED DESCRIPTION:
Objective: To evaluate the impact of the use of zinc in the prevention, incidence and severity of oral mucositis in patients with acute lymphoblastic leukemia in chemotherapy (induction and consolidation phase) of the National Institute of Pediatrics and the Federico Gómez Children's Hospital of Mexico during the period from 2019 to 2020.

Methodology: Double-blind randomized clinical trial conducted in pediatric patients with newly diagnosed or relapsed acute lymphoblastic leukemia. The subjects will be randomized to designate them in the control group (Group1 placebo) or intervention group (Group 2 zinc). The zinc / placebo intervention will be administered orally in tablets of 50-100 mg / day, from day 1 of chemotherapy until the end of the consolidation phase (2 to 2.5 months). For the detection of OM the mucositis scale of the World Health Organization will be used and the observation times will correspond to day 1, 4, 7, 14 and 21 of each chemotherapy cycle. Patients of both groups with OM will receive the same treatment (mouthwash of Gelclair) and will be observed daily until healing to determine the days of recovery.

Statistical analysis: Independent t-test and Chi-square test for the difference between the two study groups, ANOVA to compare the groups with respect to the severity of OM.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 18 years
* Patients with recent diagnosis of ALL or relapse
* Pacientes who accept by informed consent to participate in the study.

Exclusion Criteria:

* Patients with another disease or systemic condition in addition to ALL.
* Patients with Down syndrome
* Patients allergic to zinc or mannitol.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of oral mucositis | Participants will be followed for the duration of the induction and cosolidation phase of chemotherapy, an expected average of 2 to 2.5 months.
  Presence /absence The presence of oral mucositis will be measured in all patients during the induction and consolidation phase of chemotherapy.
Oral mucositis grade | Day 1 oral mucositis start to healing (1-14 days).
  World Health Organization (WHO) Criteria of Oral Mucositis The total score of this scale ranges from 0 to 4. Grade 0: no changes in the oral cavity are detected. Grade I: pain and erythema in mucosa, gums, tongue or palate. Grade II: erythema and ulcers, still with a solid diet tolerance. grade III: oral ulcers, tolerance to pasty foods and liquid diets. Grade IV: ulcers, erythema, pain, inability to swallow fluids, impossible oral feeding, and narcotic requirement to relieve pain.
Pain intensity: Visual analog scale | Day 1 oral mucositis start to healing (1-14 days).
  Visual analog scale Analogous visual scale of facial expressions, which is used in children 3 years and older. It is made up of faces with different expressions that represent a person who is happy because they do not feel pain or who is sad because they feel some pain or a lot of pain. A score is assigned to each face. The patient is asked to select the face that best describes how he feels.
  It will be recorded by the numerical score and will then be coded as follows:
  0-2 No pain 3-4 Mild 5-6 Moderate 7-8 Intense 9-10 Maximum

SECONDARY OUTCOMES:
Presence of opportunistic oral infections | Day 1, 4, 7, 14 and 21 of the induction and consolidation phase.
  Clinical or laboratory test. Record of suggestive lesions by C. albicans and determination by means of KOH, suggestive lesions of herpes and determination by PCR, suggestive bacterial lesions and detection through cultures.
  0. Absent
  1. Fungal
  2. Bacterial
  3. Viral
Neutropenia | During the induction and consolidation phase. Day 1, 4, 7, 14 and 21 of each phase. (2 to 2.5 months)
  Absolute neutrophil count obtained by laboratory test (blood count).
  0. Absence of neutropenia
  1. Mild: 1,000-1,500 / ml
  2. Moderate: 500-1,000 / ml
  3. Severe: <500 / ml

CONTACTS AND LOCATIONS:
Overall Officials: Marta M Zapata, Doctor, Principal Investigator — National Institute of Pediatrics; Luis E Juárez, Doctor, Principal Investigator — Federico Gomez Children's Hospital of Mexico
Locations (1):
- Marta M. Zapta Tarrés, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowal KA, Alaizari NA, Tarakji B, Petro W, Hussain KA, Altamimi MA. DENTAL CONSIDERATIONS FOR LEUKEMIC PEDIATRIC PATIENTS: AN UPDATED REVIEW FOR GENERAL DENTAL PRACTITIONER. Mater Sociomed. 2015 Oct;27(5):359-62. doi: 10.5455/msm.2015.27.359-362. Epub 2015 Oct 5. PMID 26622207
- [Background] Tian X, Chen WQ, Liu XL, Pi YP, Chen H. Efficacy and safety of oral zinc sulfate in the prevention of chemotherapy-induced oral mucositis: Protocol for a meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 May;97(21):e10839. doi: 10.1097/MD.0000000000010839. PMID 29794779
- [Background] Rambod M, Pasyar N, Ramzi M. The effect of zinc sulfate on prevention, incidence, and severity of mucositis in leukemia patients undergoing chemotherapy. Eur J Oncol Nurs. 2018 Apr;33:14-21. doi: 10.1016/j.ejon.2018.01.007. Epub 2018 Feb 2. PMID 29551172
- [Background] Miller MM, Donald DV, Hagemann TM. Prevention and treatment of oral mucositis in children with cancer. J Pediatr Pharmacol Ther. 2012 Oct;17(4):340-50. doi: 10.5863/1551-6776-17.4.340. PMID 23413048
- [Background] He M, Zhang B, Shen N, Wu N, Sun J. A systematic review and meta-analysis of the effect of low-level laser therapy (LLLT) on chemotherapy-induced oral mucositis in pediatric and young patients. Eur J Pediatr. 2018 Jan;177(1):7-17. doi: 10.1007/s00431-017-3043-4. Epub 2017 Nov 11. PMID 29128883
- [Background] Sangthawan D, Phungrassami T, Sinkitjarurnchai W. A randomized double-blind, placebo-controlled trial of zinc sulfate supplementation for alleviation of radiation-induced oral mucositis and pharyngitis in head and neck cancer patients. J Med Assoc Thai. 2013 Jan;96(1):69-76. PMID 23720981
- [Background] Mehdipour M, Taghavi Zenoz A, Asvadi Kermani I, Hosseinpour A. A comparison between zinc sulfate and chlorhexidine gluconate mouthwashes in the prevention of chemotherapy-induced oral mucositis. Daru. 2011;19(1):71-3. PMID 22615642
- [Background] Hayashi H, Kobayashi R, Suzuki A, Yamada Y, Ishida M, Shakui T, Kitagawa J, Hayashi H, Sugiyama T, Takeuchi H, Tsurumi H, Itoh Y. Preparation and clinical evaluation of a novel lozenge containing polaprezinc, a zinc-L-carnosine, for prevention of oral mucositis in patients with hematological cancer who received high-dose chemotherapy. Med Oncol. 2016 Aug;33(8):91. doi: 10.1007/s12032-016-0795-z. Epub 2016 Jul 14. PMID 27418192
- [Background] Arbabi-kalati F, Arbabi-kalati F, Deghatipour M, Ansari Moghadam A. Evaluation of the efficacy of zinc sulfate in the prevention of chemotherapy-induced mucositis: a double-blind randomized clinical trial. Arch Iran Med. 2012 Jul;15(7):413-7. PMID 22724877
- [Background] Mansouri A, Hadjibabaie M, Iravani M, Shamshiri AR, Hayatshahi A, Javadi MR, Khoee SH, Alimoghaddam K, Ghavamzadeh A. The effect of zinc sulfate in the prevention of high-dose chemotherapy-induced mucositis: a double-blind, randomized, placebo-controlled study. Hematol Oncol. 2012 Mar;30(1):22-6. doi: 10.1002/hon.999. Epub 2011 Jun 21. PMID 21692101

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT04321850/Prot_SAP_ICF_000.pdf